CLINICAL TRIAL: NCT04299165
Title: Impact of a Smartphone Application (KAIA COPD-App) in Combination With Activity Monitoring as Maintenance Program Following Pulmonary Rehabilitation in COPD: an International Multi-centered Randomized Controlled Trial
Brief Title: Smartphone-App as Maintenance Program in COPD
Acronym: AMOPUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaia Health Software (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kaia COPD 001; DRKS00017275 (Registry Identifier: DRKS)
Record Dates: First submitted 2020-02-19; First posted 2020-03-06 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; COPD; Medical Mobile application; Digital Therapeutics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device: KAIA COPD-App (Medical Mobile Application). (Experimental): The study intervention is an exercise training program that requires only a chair or water bottles, consisting of training elements with progressive levels of intensity, individually adaptable to the participant's exercise level. This training program is delivered to the participants with the help of KAIA COPD-App. Additionally, the Polar A370 watch will collect the daily symptoms and training log during each session for the Database.
  Interventions: Device: Kaia COPD Application
- Usual Care (Active Comparator): The Training of the control-group is performed by regular recommendations/ Standard of care. Standard of care in this context means to hand out the brochure " Besser Leben mit COPD " including an emergency plan, providing exercise training examples, to hand out addresses of out-patient physiotherapists and to hand out a detailed medical report including medical recommendations.Additionally, the Polar A370 watch will collect the daily symptoms and training log during each session for the Database.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Kaia COPD Application — The study intervention consists of training sessions conducted daily by the patient via the COPD-App.
  Arms: Device: KAIA COPD-App (Medical Mobile Application).
Other: Usual Care — The control group will also be an active control as participants receive a leaflet to convey an active lifestyle and a list of exercises to do at home.
  Arms: Usual Care

SUMMARY:
Increasing Physical activity (PA) is considered to be an important factor in an efficient management of the chronic obstructive pulmonary disease (COPD). The successful methods required to achieve improvements in PA following Pulmonary Rehabilitation (PR), however are sparsely reported. Therefore, the investigators conduct this trial to evaluate the effectiveness of using a COPD management program delivered to the patient through a mobile medical application Kaia COPD-App, after the completion of a PR.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multi-centered trial carried out at in-patient PR-hospital centers in Germany and Switzerland . The interventions will involve use of KAIA COPD-app program (Arm 1) or an active comparator i.e. usual care (Arm 2). Patients completing an in-hospital PR-Program and consenting to participate in the study will be screened for the inclusion and exclusion criteria and enrolled in the study. After fulfillment of the screening requirements, they will be randomized into one of the two arms with parallel group assignment in a 1:1 ratio. The training program will be delivered to the participants grouped to the arm 1 through KAIA COPD-App and arm 2 as provided in regular recommendations or standard of care through the PI. In total, 104 participants will be included to the trial. Treatment period will last for 24 weeks. Electronic versions of Questionnaires will be used to collect patient reported assessments remotely. The primary outcome measure is the change in physical activity of the intervention group in comparison to the control group, measured over one week as mean steps per day with the Polar A 370 activity tracker, from baseline (end of PR) to 6-months follow-up. The secondary outcome measures are functional exercise capacity, health status, sleep quality, exacerbation rate, depression and anxiety symptoms assessed at several intervals.

This study seeks to prove the implications of the Kaia COPD mobile application in COPD patients after PR. The app offers educational, exercise training plus activity monitoring and motivational program that can be easily implemented in the patient's home-setting enabling patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD Patients willing and able to sign informed consent for use of their pseudonymized clinical data within the scope of the present interventional trial
* COPD patients who have completed an in-hospital pulmonary rehabilitation program with an average duration of 2-3 weeks.
* Diagnosis of COPD, defined as forced expiratory volume in 1s/forced vital capacity (FEV1/FVC) <70% predicted, FEV1<80 % predicted after bronchodilation, with or without chronic symptoms (cough, sputum production) corresponding to a GOLD stage II-IV
* Completion of the screening period and fulfilling of the randomization criteria as defined by the protocol
* Ability to use a smartphone and smartphone-apps
* Willingness to wear an activity tracker during study period of 6 months
* Patients ≥40 years of age.
* Knowledge of German language to understand study material, assessments and contents of the COPD-App

Exclusion Criteria:

* The Patient is not able to conduct the exercise training program due to physical, cognitive or safety reasons, as judged by investigator; e.g., lower limb joint surgery within preceding 3 months, unstable cardiac disease, predominant neurological limitations, planned surgical or other interventions disturbing the study intervention.
* Significant psychiatric disorders, legal incapacity or limited legal capacity.
* Patients participation in another clinical trial with an investigational medication within 30 days prior to study entry.
* Patients already using the KAIA COPD App

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
Steps per day as mean over one week from baseline until the treatment end | Every day for 6 months
  The primary outcome are the steps per day as mean over one week from baseline (second week after discharge from PR) to 6 months follow-up in the intervention group in comparison to the control group as an equivalent for the physical activity of the participants, measured by an activity tracker (Polar A370-Watch).

SECONDARY OUTCOMES:
Dyspnea | Baseline, Visit 5 (12 weeks) and Visit 8( 24 weeks)
  Dyspnea will be assessed by the COPD Assessment Test (CAT) which measures the impact of COPD on a person's health status (8 questions, 6-point Likert-type scale)
Functional exercise capacity using I min Sit to stand test | Baseline (day 0), Visit 5 (12 weeks) and Visit 8( 24 weeks)
  Functional exercise capacity will be assessed by the widely-used and validated 1-min sit-to-stand test (STS). The patients are guided through an integrated video with a stop watch in an ePRO to perform the test in a right way in home settings.
Quality of life through SAS-CRQ | Baseline (day 0), Visit 5 (12 weeks) and Visit 8( 24 weeks)
  SAS- CRQ The chronic respiratory questionnaire, a self-administered instrument, includes 20 items across four domains: dyspnea (5 items), fatigue (4 items), emotional function (7 items), and mastery (4 items). Patients will be scored for the Quality of life around their experience on a 7-point scale ranging from 1 (maximum impairment) to 7 (no impairment).
Subjective health status | At the Baseline (Day 0) and every 4 weeks (V2 to V8) until the end of treatment period of 24 weeks
  A feeling thermometer scale allows respondents to rank how positively individuals feels about the quality of life to measure individuals' subjective health status. The scale ranges from a minimum of 0 to a maximum of 100.
Sleep efficacy and total sleep time | Every night for 6 months of treatment period
  Sleep efficacy (SE) and total sleep time (TST)will be measured by the Polar A370 Watch every night during the treatment period.
Motivation for reaching his or her individual defined goal of physical activity | At the Baseline (Day 0) and every 4 weeks (V2 to V8) until the end of treatment period of 24 weeks
  This assessment is linked to the intervention group using COPD App only. During monthly visits, a certain number of steps will be fixed as a goal for the patients in the COPD application.
Assessment of usability | End of the treatment period of 24 weeks from baseline
  This assessment is linked to the intervention group using COPD App only. The use of the application will be assessed every week through patient data reports captured in the COPD Application.
Rate, number and severity of adverse events | At baseline (day 0) and every 2 weeks after, until the end of the treatment period of 24 weeks
  The AEs and SAEs will be documented to assess the safety related to the use of the application and trainings, in the home settings.
Rate, number and severity of device deficiencies | At baseline(day 0) and every 2 weeks after, until the end of the treatment period of 24 weeks
  The DDs will be documented to assess the performance of the device and usability.
Hospital Anxiety and Depression Scale | Baseline (day 0), Visit 5 (12 weeks) and Visit 8( 24 weeks)
  The HADS Questionnaire will be used to measure anxiety and depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Spielmanns, MD, Principal Investigator — Reha Zentrum Wald, Zürich
Locations (2):
- Koczulla, Schönau am Königssee, Germany
- Zürcher RehaZentren Wald, Wald, Switzerland

IPD SHARING:
Plan to Share IPD: No